CLINICAL TRIAL: NCT07224074
Title: Impact of Exogenous Ketones on Sleep and Breathing in Healthy Volunteers (K-EFFECTS)
Brief Title: Impact of Exogenous Ketones on Sleep and Breathing in Healthy Volunteers (K-SLEEP)
Acronym: K-SLEEP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: HVMN Inc (Industry); KETONE-IQ (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00517978
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Sleep
Keywords: Sleep; Healthy; Ketones
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: All participants will take open-label Ketone IQ before bedtime at two different doses (20 or 40 g).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- K-SLEEP (Experimental): Healthy Participants will ingest (1) Ketone IQ 20 g or (2) Ketone IQ 40 g before bedtime and undergo objective and subjective sleep assessments.
  Interventions: Dietary Supplement: KETONE-IQ 20 grams (g); Dietary Supplement: KETONE-IQ 40 grams (g)

INTERVENTIONS:
Dietary Supplement: KETONE-IQ 20 grams (g) — Dietary Supplement: Ketone-IQ (1,3 Butanediol) Description: Ketone-IQ (1,3 Butanediol) 20g will be ingested (open-label) before bedtime.
Dietary Supplement: KETONE-IQ 40 grams (g) — Dietary Supplement: Ketone-IQ (1,3 Butanediol) Description: Ketone-IQ (1,3 Butanediol) 40g will be ingested (open-label) before bedtime.

SUMMARY:
Ketones are molecules generated by the body during the metabolism of fat. Exogenous ketones (EK) are substances that can raise the level of ketones in the circulation without changing diet. In this research study, the investigators are testing the tolerability, sleep effects, and dose effects of a commercially available EK product called Ketone-IQ.

The investigators will administer Ketone-IQ open-label to healthy volunteers (n=20, 10 men, 10 women) before sleep in the participant's home setting and collect information about subjective sleep and GI symptoms, as well as objective data about beta-hydroxybutyrate (BHB) levels and sleep architecture using a headband-EEG device (Sleep Profiler). Participants will measure capillary BHB levels before ingestion and at 1, 3, and 5 hours post-ingestion, as well as upon awakening.

Questionnaires will be used to gather feedback on the palatability of EK, GI side effects, and sleep quality. Higher scores indicate better sleep quality. Two doses (20 g and 40 g) of Ketone-IQ will be tested each for two nights, with one night used to measure BHB levels and a separate night to allow for uninterrupted sleep.

DETAILED DESCRIPTION:
There is growing interest leveraging ketone metabolism for human health and performance. Exogenous ketones (EK) are substances that directly increase circulating ketones in the body without requiring a change in diet. While EK have been studied in the contexts of energy metabolism and exercise, few studies have examined EKs impact on sleep, a critical window for repair and rest. A mouse study showed that wakefulness increased brain ketones, while injection of acetoacetate increased slow wave sleep, suggesting a homeostatic sleep-promoting role of ketones. In humans, strenuous exercise reduced rapid eye movement (REM) sleep, which was prevented by ingestion of a ketone ester before sleep. Otherwise, few studies have systematically evaluated the effects of EK on sleep architecture and quality.

To examine the potential of EK to affect sleep, the investigators are conducting the K-SLEEP study. The investigators will examine sleep architecture and quality and BHB levels when EK are ingested prior to sleep (n=20). Healthy volunteers will ingest EK or placebo 30 minutes before sleep. Participants will measure capillary BHB levels before ingestion and at 1, 3, 5, hours post-ingestion as well as upon awakening. Questionnaires will solicit feedback about EK palatability, GI side effects, and sleep quality. Two doses will be examined, 20 g or 40 g with 1-2 days of washout between doses.

EK come in several forms including 1,3BD, ketone esters (beta-hydroxybutyrate + 1,3BD), fatty acid esters (C6 or C8 medium chain fatty acids + 1,3 BD), free acid ketones (beta-hydroxybutyric acid), and ketone salts (combination of ketone body with a mineral salt such as sodium or potassium). 1,3BD can be ingested in isolation or in a combination formulation (5, 6) whereupon it is absorbed and converted by hepatic enzymes into gamma-hydroxybutyrate and then oxidized to the ketone body BHB. In this study, the investigators will utilize a commercially available formulation of 1,3BD called Ketone IQ. This product has a more gradual onset and prolonged period of ketosis than ketone salt ingestion, making it more suitable for inducing sustained ketosis during several hours of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years old with a BMI of 18 - 30 kg/m^2

Exclusion Criteria:

* No concomitant sleep disorder (e.g. sleep apnea, insomnia, restless leg syndrome, narcolepsy, idiopathic hypersomnia). If there is no known diagnosis of sleep apnea, a STOP-BANG score of 5 or higher is an exclusion.
* No current daytime respiratory impairment such as uncontrolled asthma, or uncontrolled Chronic Obstructive Pulmonary Disease (COPD), pneumonia, interstitial lung disease.
* No known history of chronic renal disease or diabetes (type 1 or type 2).
* No use of supplemental oxygen.
* Cannot be on a low carbohydrate (<130 g carbohydrate/day) or ketogenic diet, intermittent fasting, or consuming exogenous ketones
* Cannot be pregnancy or breastfeeding
* Cannot be on medications: acetazolamide or Sodium-glucose cotransporter-2 (SGLT2) inhibitor (10), daily opioid use.
* K-BREATHE: no history of claustrophobia or panic disorder
* Frequent alcohol intake (more than 1 drink per day on average, or > 10 drinks per week).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Beta hydroxybutyrate (BHB) maximal concentration (Cmax) | 1, 3, 5 hours, and final awakening (Night 2); and 1, 3, 5 hours, and final awakening (Night 5)
  Participants will measure their capillary BHB levels at home at 4 time points after ingestion (1, 3, 5 hours, and final awakening). The investigators will derive the maximal BHB concentration (mmol) of these timepoints. Measured on two occasions: Night 2 (Ketone IQ 20 g) and Night 5 (Ketone IQ 40 g).

SECONDARY OUTCOMES:
Sleep quality as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance (SD) short from 8a | day 2, day 4, and day 7
  Modified PROMIS-SD short form 8a: Uses a Likert-type response scale. The raw score range is 8 to 40 with a higher score indicating greater severity of sleep disturbance.
Sleep quality as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment (SRI) short form 8a | day 2, day 4, and day 7.
  Modified PROMIS-SRI short form 8a: uses a Likert-type response scale. The raw score range is 8 to 40 with a higher score indicating greater severity of sleep related impairment.
Sleep quality as assessed by Stanford Sleepiness Scale | 3 questionnaires in 1 week on day 2, day 4, and day 7.
  Stanford Sleepiness Scale; Total score range: 0-7. 7 Sleep quality 7 being the worst
Sleep architecture as assessed by minutes of sleep in each stage | Night 1, Night 2, Night 3, Night 6
  Measured using a Sleep Profiler device, the Sleep Profiler provides automated sleep staging validated against polysomnography (PSG), using EEG signals to quantify time spent in each sleep stage. Worn for about 8 hours each night.
Gastrointestinal tolerability as assessed by the Gastrointestinal Symptoms Questionnaire | day 3, day 4, day 6, and day 7
  Questionnaire about GI tolerability of product; 0-8, 8 being "unbearable"

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided at publication, accompanied by a data dictionary, and preserved for at least five years. De-identified experimental data, including sleep data, questionnaires, and BHB measurements may be shared by the PI upon reasonable requested.
Supporting Information: Study Protocol
Time Frame: Deidentified scientific data included in published manuscripts will be made available at the time of publication, and additional data will be made available to researchers upon request. Data will be made available for up to 3 years following study completion.
Access Criteria: To request access to the data, researchers will be able to contact Dr. Jonathan Jun via email. Any data attached as a supplement to publications will be available for download from the publisher's website. The intention is to allow qualified external investigators broad access to the study data for specified research purposes.